CLINICAL TRIAL: NCT06177457
Title: A PHASE 1, MULTI-PART RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO CONTROLLED STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF MULTIPLE ASCENDING ORAL DOSES OF PF-07293893 IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Understand the Effect of Multiple Ascending Doses of PF-07293893 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: C5171002; 2023-508171-36-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Healthy Participants
Keywords: PF-07293893; Multiple ascending dose; Safety; Tolerability; Pharmacokinetics
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- PF-07293893 and Placebo (Cohort 1) (Experimental): Dose level 1: Multiple dose administration of PF-07293893 and placebo over 14 days in healthy participants; 6 participants will receive PF-07293893 and 2 will receive placebo.
  Interventions: Drug: PF-07293893; Drug: Placebo
- PF-07293893 and Placebo (Cohort 2) (Experimental): Dose level 2: Multiple dose administration of PF-07293893 and placebo over 14 days in healthy participants; 6 participants will receive PF-07293893 and 2 will receive placebo.
  Interventions: Drug: PF-07293893; Drug: Placebo
- PF-07293893 and Placebo (Cohort 3) (Experimental): Dose level 3: Multiple dose administration of PF-07293893 and placebo over 14 days in healthy participants; 6 participants will receive PF-07293893 and 2 will receive placebo.
  Interventions: Drug: PF-07293893; Drug: Placebo
- PF-07293893 and Placebo (Cohort 4) (Experimental): Dose level 4: Multiple dose administration of PF-07293893 and placebo over 14 days in healthy participants; 6 participants will receive PF-07293893 and 2 will receive placebo.
  Interventions: Drug: PF-07293893; Drug: Placebo
- PF-07293893 and Placebo (Cohort 5) (Experimental): Dose level 5: Multiple dose administration of PF-07293893 and placebo over 14 days in healthy participants; 6 participants will receive PF-07293893 and 2 will receive placebo.
  Interventions: Drug: PF-07293893; Drug: Placebo
- PF-07293893 and Placebo (Cohort 6, Optional) (Experimental): Dose level 6: Multiple dose administration of PF-07293893 and placebo over 14 days in healthy participants; 6 participants will receive PF-07293893 and 2 will receive placebo.
  Interventions: Drug: PF-07293893; Drug: Placebo
- Midazolam drug-drug interaction (Cohort 7, Optional) (Experimental): Drug-drug interaction assessment of pharmacokinetics interaction in PF-07293893 and midazolam
  Interventions: Drug: PF-07293893; Drug: Midazolam
- Metabolism and elimination of PF-07293893 (Cohort 8, Optional) (Experimental): Determination of excretion routes and metabolite profiling of PF-07293893.
  Interventions: Drug: PF-07293893
- Skeletal muscle imaging (Cohort 8, optional) (Experimental): Evaluation of the effect of 14-days of daily PF-07293893 on skeletal muscle glycogen in healthy adult participants
  Interventions: Drug: PF-07293893; Drug: Placebo

INTERVENTIONS:
Drug: PF-07293893 — PF-07293893 will be administered as tablets every day (QD) over 14 days
Drug: Placebo — Placebo will be administered as tablets; QD over 14 days
  Arms: PF-07293893 and Placebo (Cohort 1); PF-07293893 and Placebo (Cohort 2); PF-07293893 and Placebo (Cohort 3); PF-07293893 and Placebo (Cohort 4); PF-07293893 and Placebo (Cohort 5); PF-07293893 and Placebo (Cohort 6, Optional); Skeletal muscle imaging (Cohort 8, optional)
Drug: Midazolam — Single doses of Midazolam will be administered as oral solution alone and in combination with PF-07293893
  Arms: Midazolam drug-drug interaction (Cohort 7, Optional)

SUMMARY:
This study has four parts: Part A, Part B, Part C, and Part D.

The purpose of Part A of this study is to learn about the:

* safety,
* tolerability,
* how PF-07293893 is processed by the body when multiple doses of PF-07293893 are given to healthy participants.

The purpose of Part B of this study is to understand the effect of multiple doses of PF-07393893 on the amount of midazolam when given as a single dose by mouth.

The purpose of part C of this study is to understand how PF-07293893 is changed in the body and how much PF-07293893 and it's changed forms are being removed in urine and feces after a single dose given to single participants.

The purpose of Part D is to understand the effect of multiple doses of PF-07293893 on the amount of glycogen (storage form of glucose) in the muscle of healthy participants.

Part B, C and D will be done if the results of Part A support further study of PF-07293893.

The study is seeking participants who:

* are females who are not able to give birth to a child. These female participants should be between 18 to 65 years of age.
* are males of 18 to 65 years of age.
* have a body mass index (BMI) of 20.0 to 35.0 kilograms per squared meter.
* have total body weight of more than 45 kilograms (99 pounds).

For a given participant in Part A, the total study is going to last up to about 11 weeks. This includes from the time of selection till the last follow-up phone call. The participants will be selected if they are fit for the study 28 days before the first dose of the study medicines. Participants who are selected will be admitted to the study site on Day 1 for around 18 days. Following discharge, participants will return for an on-site follow-up visit 7 to 10 days after receiving the final dose of the study medicine. The follow-up contact may be via a telephone call and will happen 28 to 35 days after the final dose of study medicine is given.

For a given participant in Part B, the total study is going to last up to about 11 weeks. This study consists of 4 periods. Participants will be admitted to the study site on Day 1 and discharged on Day 3 in period 4. Following discharge, participants will return for an on-site follow-up visit 7 to 10 days after receiving the final dose of the study medicine in period 4. The follow-up contact may be via a telephone call and will happen 28 to 35 days after the final dose of study medicine is given in period 4.

For a given participant in Part C, the total study is going to last up to about 9 weeks. Participants will be admitted to the study site on Day 1. The participants will be discharged on Day 11 after giving the study medicine. The follow-up contact may be via a telephone call and will happen 28 to 35 days after the final dose of study medicine is given.

For a given participant in Part D, the total study is going to last up to about 11 weeks. The participants will be selected if they are fit for the study 28 days before the first dose of the study medicines. Participants who are selected will be admitted to the study site on Day -3 for around 17 days. Following discharge, participants will return for an on-site follow-up visit 7 to 10 days after receiving the final dose of the study medicine. The follow-up contact may be via a telephone call and will happen 28 to 35 days after the final dose of study medicine is given.

ELIGIBILITY:
Inclusion Criteria:

* Females of non-childbearing potential and males 18 to 65 years of age (except for optional Part C in which only males will be recruited), inclusive, at the time of signing the ICD who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* BMI of 20-35 kg/m2; and a total body weight >45kg (99 lb).
* Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures. Capable of giving signed informed consent.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, ophthalmologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).

History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed.

* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Part C Only: History of irregular bowel movements including irritable bowel syndrome or frequent episodes of diarrhea or constipation defined by less than 1 bowel movement on average per 2 days or lactose intolerance.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention with the exception of moderate/strong CYP3A inducers or inhibitors which are prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention.
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during their participation in this study.
* Previous exposure to PF-07293893 treatment.
* A positive urine drug test.
* Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm/Hg for participants ≥60 years old, following at least 5 minutes of supine rest. If systolic BP is ≥ 140 or 150 mm Hg (based on age) or diastolic ≥90 mm Hg, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
* Renal impairment as defined by an estimated glomerular filtration rate (eGFR) <75 mL/min/1.73m². Since participants are 18 years to 65 years, 2021 Screat-based CKD-EPI eGFR is the recommended formula.
* Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete LBBB, signs of an acute or indeterminate- age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third- degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If QTcF exceeds 450 ms, or QRS exceeds 120 ms, the ECG should be repeated twice and the average of the 3 QTcF or QRS values used to determine the participant's eligibility. Computer interpreted- ECGs should be overread by a physician experienced in reading ECGs before excluding a participant.
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study -specific laboratory and confirmed by a single repeat test, if deemed necessary: ALT, AST, Bili ≥ 1.05 x ULN. participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.

CK > 2.5 x ULN.

* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit, or 3 ounces (90 mL) of wine).
* Use of tobacco or nicotine-containing products in excess of the equivalent of 5 cigarettes/day or 2 chews of tobacco/day.
* Part B Only: History of sensitivity reaction to midazolam, or any of the formulation components.
* Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.
* Part D Only: Any contra-indication to Magnetic Resonance Imaging, including noncompatible metallic implants, severe claustrophobia, or the inability to remain still for the duration of the scan session.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Part A:Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline up to 35 days after last dose of study intervention (approximately 11 weeks).
Part A: Number of Participants With Clinical Laboratory Abnormalities | Baseline up to 10 days after last dose of study intervention (approximately 7 weeks).
Part A: Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to 10 days after last dose of study intervention (approximately 7 weeks).
Part A: Number of Participants With Change From Baseline in Electrocardiogram (ECG) Findings | Baseline up to 10 days after last dose of study intervention (approximately 7 weeks).
Part A: Number of Participants With Clinically-Significant Change From Baseline in Physical Examination Findings | Baseline up to 10 days after last dose of study intervention (approximately 7 weeks).
Part A: Number of Participants With Clinically-Significant Change From Baseline in Neurological Examination Findings | Baseline up to 10 days after last dose of study intervention (approximately 7 weeks).
Part B: Maximum Observed Plasma Concentration (Cmax) of Midazolam | Time Frame: predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16 and 24 hours post dose on Period 1/Day 1
Part B: Maximum Observed Plasma Concentration (Cmax) of Midazolam | Time Frame: predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 and 36 hours post dose on Period 2/Day 2
Part B: Maximum Observed Plasma Concentration (Cmax) of Midazolam | Time Frame: predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post dose on Period 4/Day 1
Part B: Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUClast) of Midazolam | Time Frame: predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16 and 24 hours post dose on Period 1/Day 1
Part B: Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUClast) of Midazolam | Time Frame: predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 and 36 hours post dose on Period 2/Day 2
Part B: Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUClast) of Midazolam | Time Frame: predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post dose on Period 4/Day 1
Part B: Area under the plasma concentration-time curve from time 0 to Extrapolated Infinite Time (AUCinf) of Midazolam | Time Frame: predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16 and 24 hours post dose on Period 1/Day 1
Part B: Area under the plasma concentration-time curve from time 0 to Extrapolated Infinite Time (AUCinf) of Midazolam | Time Frame: predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 and 36 hours post dose on Period 2/Day 2
Part B: Area under the plasma concentration-time curve from time 0 to Extrapolated Infinite Time (AUCinf) of Midazolam | Time Frame: predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post dose on Period 4/Day 1
Part C: Total recovery of drug-related material in urine and feces separately, and both routes combined, expressed as a percent of total dose administered. | Predose to Day 11
Part D: Change from baseline in glycogen on Day 14 as measured by 13C MRS of skeletal muscle | Day 14 (last day of dosing)

SECONDARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of PF-07293893 | predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24 hours post dose on Day 1
Part A: Maximum Observed Plasma Concentration (Cmax) of PF-07293893 | predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post dose on Day 14
Part A: Area Under the Plasma Concentration-Time Curve From Time 0 to Dosing Interval (tau) (AUCtau) of PF-07293893 | predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24 hours post dose on Day 1
Part A: Area Under the Plasma Concentration-Time Curve From Time 0 to Dosing Interval (tau) (AUCtau) of PF-07293893 | predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post dose on Day 14
Part A: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-07293893 | predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24 hours post dose on Day 1
Part A: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-07293893 | predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post dose on Day 14
Part A: Amount of PF-07293893 Excreted Unchanged in Urine Over the Dosing Interval Tau (Aetau) | On Day 14, urine collection for PK to occur over 0-tau, according to dosing frequency (ie, 0-12 hours for 12 hour dosing interval; 0-24 hours for 24 hour dosing interval)
Part A: Percentage of Dose of PF-07293893 Excreted Unchanged in the Urine Over the Dosing Interval Tau (Aetau%) | On Day 14, urine collection for PK to occur over 0-tau, according to dosing frequency (ie, 0-12 hours for 12 hour dosing interval; 0-24 hours for 24 hour dosing interval)
Part A: Renal Clearance of PF-07293893 | On Day 14, urine collection for PK to occur over 0-tau, according to dosing frequency (ie, 0-12 hours for 12 hour dosing interval; 0-24 hours for QD dosing interval)
Part B: Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline up to 35 days after last dose of study intervention (approximately 10 weeks)
Part B: Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to 10 days after last dose of study intervention (approximately 7 weeks)
Part B: Number of Participants With Change From Baseline in Electrocardiogram (ECG) Findings | Baseline up to 10 days after last dose of study intervention (approximately 7 weeks)
Part B: Number of Participants With Clinical Laboratory Abnormalities | Baseline up to 10 days after last dose of study intervention (approximately 7 weeks)
Part B: Number of Participants With Clinically-Significant Change From Baseline in Physical Examination Findings | Baseline up to 35 days after last dose of study intervention (approximately 10 weeks)
Part C: Maximum Observed Plasma Concentration (Cmax) of PF-07293893 | predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 hours post dose
Part C: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-07293893 | predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 hours post dose
Part C: Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUClast) of PF-07293893 | predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 hours post dose
Part C: Area under the plasma concentration-time curve from time 0 to Extrapolated Infinite Time (AUCinf) of PF-07293893 | predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 hours post dose
Part C: Terminal half life (t1/2) of PF-07293893 | predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 hours post dose
Part C: Apparent clearance (CL/F) of PF-07293893 from plasma | predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 hours post dose
Part C: Apparent volume of distribution (Vz/F) of PF-07293893 | predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 hours post dose
Part D: Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline up to 35 days after last dose of study intervention (approximately 11 weeks)
Part D: Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to 10 days after last dose of study intervention (approximately 8 weeks)
Part D: Number of Participants With Change From Baseline in Electrocardiogram (ECG) Findings | Baseline up to 10 days after last dose of study intervention (approximately 8 weeks)
Part D: Number of Participants With Clinical Laboratory Abnormalities | Baseline up to 10 days after last dose of study intervention (approximately 8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (2):
  - Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut
  - Yale University/Magnetic Resonance Research Center (MRRC), New Haven, Connecticut
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5171002